CLINICAL TRIAL: NCT01414751
Title: Interventions for Chronic Diseases: Effect of Patient Values and Effectiveness Information on Patients' Choice of Therapy, Adherence to Therapy and Satisfaction With Therapy
Brief Title: Influence of Intervention Methodologies on Patient Choice of Therapy
Acronym: IMPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Charlotte Gry Harmsen, MD PhD fellow, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CGH001
Record Dates: First submitted 2011-08-05; First posted 2011-08-11 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Communication; Hypercholesterolemia
Keywords: Risk communication; Shared decision making; Cardiovascular diseases; Hypercholesterolemia; Prevention
MeSH Terms: conditions — Communication; Hypercholesterolemia; Cardiovascular Diseases | interventions — Numbers Needed To Treat; Life Support Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Absolute risk reduction information (Active Comparator): Patients belonging to this arm receive effectiveness information by means of absolute risk reduction when talking with their general practitioner concerning their cholesterol level and possible gain if starting therapy.
  Interventions: Behavioral: Absolute risk reduction
- Prolongation of life information (Active Comparator): Patients belonging to this arm receive effectiveness information by means of prolongation of life/life extension when talking with their general practitioner concerning their cholesterol level and possible gain if starting therapy.
  Interventions: Behavioral: Prolongation of life

INTERVENTIONS:
Behavioral: Absolute risk reduction — Patients receive effectiveness information concerning cholesterol lowering therapy by means of absolute risk reduction
  Other Names: ARR
  Arms: Absolute risk reduction information
Behavioral: Prolongation of life — Patients receive effectiveness information concerning cholesterol lowering therapy by means of prolongation of life/life extension.
  Other Names: POL
  Arms: Prolongation of life information

SUMMARY:
Few studies have explored how specific formats of effectiveness information effect on real patients' decisions. We only know little about what kind of format would be the optimal to help patients make well-informed real-life decisions corresponding to their preferences.

The trial is developed in a clinical randomised design to study risk communication in the shared decision making between general practitioners (GP) and their patients in primary prevention with of cholesterol lowering drug. Endpoints are effect of GPs' information about treatment effectiveness and their patients' values on patients' tendency to accept and adhere to the treatment as well as their feeling of content with the choice made. GPs are randomised to inform about risk and treatment effectiveness by means of either absolute risk reduction (ARR) or Prolongation of Life (POL). Afterwards patients are invited to answer questionnaires concerning their content with decisions and reflections. Patients' redemption of prescriptions during the following week and the first year are recorded through an electronic database.

57 GPs and 248 patients have been enrolled in the trial.

DETAILED DESCRIPTION:
As chronic diseases are steadily increasing in the industrialized countries, there is a growing focus on preventive initiatives. This means that risk communication between the physician and his patients plays a central role.

Effective risk communication can enhance knowledge, involvement in decisions about tests or treatment, autonomy and empowerment of patients. Poor communication, however, can lead to anxiety, lack of confidence in health care professionals, and other adverse outcomes. It is vital that we identify the available evidence about how it should best be done.

The standard formats used to communicate intervention effectiveness are absolute risk reduction, relative risk reduction, number needed to treat, and life prolongation of life.

Few studies have explored the formats' influence on real patient decisions, implying that we only know little about what kind of format would be the optimal to help patients make well-informed real-life decisions corresponding to their preferences.

In a clinical randomized design risk communication is studied in the preventive talk between the general practitioner (GP) and his patients concerning cardiovascular diseases. Special focus is on influence of information format on patients' choice of therapy, adherence to therapy and satisfaction with therapy.

GPs are randomized to one of two groups, being taught in informing their patients by means of either absolute risk reduction, ARR or life extension, LE.

The setting is the preventive talk in the GP's clinic. From a measured total-cholesterol the GP informs his patient about the individual risk of getting a cardiovascular disease and the possible effectiveness of a cholesterol-lowering drug. This is done by means of either ARR or LE. After the talk the patient is invited to answer a questionnaire concerning personal experience with the information given (deadline 2 weeks after the talk), and again after 3 months will receive a questionnaire concerning satisfaction with the decision made and reflections. Patients' redemption of prescriptions during the following week and the first year are recorded through Odense PharmacoEpidemiological Database, OPED. The GPs' opinions, experiences and concerns about risk communication, prevention, and usage of statins are explored by means of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 40-69 year-olds
* Patients with a measured total-cholesterol of > 4 MMol/Litre

Exclusion Criteria:

* Patients with diabetes
* Patients with known chronic cardiovascular diseases
* Patients who are already being treated with cholesterol lowering therapy
* Patients who are not familiar with the danish language

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Patient's satisfaction and confidence with the information given. | Within two weeks after receiving the information and after 3 months.
  After receiving information about effectiveness of a possible therapy, patients fill in a validated questionnaire ("COMRADE") concerning confidence and satisfaction with the information given. The questionnaire is handed out immediately after information has been given (deadline for answering being two weeks after receiving the effectuveness information), and again after three months to detect adherence with the decision made.

SECONDARY OUTCOMES:
Influence of effectiveness format on patients' consent or refusal to a therapy offer | Within the first week after receiving the information and during the following year.
  After patients have received the effectiveness information the secondary study focus will be on tendency to accept the offered therapy according to information format given. This will be studied by means of patients' redemptions of prescriptions, recorded through a pharmacoepidemilogical database, as well as background information about the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dorte E Jarbol, MD PhD, Study Director — Research Unit of General Practice, Institute of Public Health, University of Southern Denmark

REFERENCES:
- [Derived] Harmsen CG, Kristiansen IS, Larsen PV, Nexoe J, Stovring H, Gyrd-Hansen D, Nielsen JB, Edwards A, Jarbol DE. Communicating risk using absolute risk reduction or prolongation of life formats: cluster-randomised trial in general practice. Br J Gen Pract. 2014 Apr;64(621):e199-207. doi: 10.3399/bjgp14X677824. PMID 24686884
- [Derived] Harmsen CG, Jarbol DE, Nexoe J, Stovring H, Gyrd-Hansen D, Nielsen JB, Edwards A, Kristiansen IS. Impact of effectiveness information format on patient choice of therapy and satisfaction with decisions about chronic disease medication: the "Influence of intervention Methodologies on Patient Choice of Therapy (IMPACT)" cluster-randomised trial in general practice. BMC Health Serv Res. 2013 Feb 25;13:76. doi: 10.1186/1472-6963-13-76. PMID 23442351